CLINICAL TRIAL: NCT02998775
Title: A Multicenter Phase 0 Study In Healthy Subjects and Subjects With Either Hepatic Or Renal Impairment To Obtain Plasma For Assessment In Vitro Lenvatinib Protein Binding
Brief Title: Phase 0 Study in Healthy, Hepatic and Renal Impaired Subjects to Obtain Plasma for Lenvatinib Protein Binding
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: E7080-A001-010
Record Dates: First submitted 2016-12-16; First posted 2016-12-20 (Estimated); Last update posted 2018-09-07 (Actual); Status verified 2018-09

CONDITIONS: Hepatic Impairment; Renal Impairment
Keywords: in vitro protein binding; hepatic impairment; renal impairment
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (8):
- 6 participants with mild renal impairment (Other): Renal Impairment Mild: creatinine clearance, 50 to 80 milliliters per minute (mL/min)
  Interventions: Drug: Plasma Sampling
- 6 participants with moderate renal impairment (Other): Renal Impairment Moderate: creatinine clearance, 30 to 49 mL/min
  Interventions: Drug: Plasma Sampling
- 6 participants with severe renal impairment (Other): Renal Impairment Severe: creatinine clearance, 15 to 29 mL/min
  Interventions: Drug: Plasma Sampling
- 8 participants normal renal status (Other): Renal status normal as defined by creatinine clearance ≥ 81 mL/min, otherwise age, gender, and smoking characteristics matching renal-impaired participants
  Interventions: Drug: Plasma Sampling
- 6 participants with mild hepatic impairment (Other): Hepatic impairment mild: total score on the Child-Pugh classification system between 5 and 6
  Interventions: Drug: Plasma Sampling
- 6 participants with moderate hepatic impairment (Other): Hepatic impairment moderate: total score on the Child-Pugh classification system between 7 and 9
  Interventions: Drug: Plasma Sampling
- 6 participants with severe hepatic impairment (Other): Hepatic impairment severe: total score on the Child-Pugh classification system between 10 and 15
  Interventions: Drug: Plasma Sampling
- 8 participants normal hepatic status (Other): Hepatic status normal, otherwise age, gender, and smoking characteristics matching hepatic-impaired participants
  Interventions: Drug: Plasma Sampling

INTERVENTIONS:
Drug: Plasma Sampling — No lenvatinib will be administered in this study; however, plasma samples will be obtained for assessment of in vitro lenvatinib protein binding.

SUMMARY:
E7080-A001-010 is a multicenter, parallel-group study in participants with mild, moderate, or severe hepatic or renal impairment and age-, gender-, and smoking status-matched healthy participants. The primary objective of the study is to obtain plasma from participants for use in in vitro protein binding studies.

DETAILED DESCRIPTION:
E7080-A001-010 is a multicenter, parallel-group study in participants with mild, moderate, or severe hepatic or renal impairment and age-, gender-, and smoking status-matched healthy participants. Approximately 6 participants with each degree (mild, moderate, or severe) of hepatic or renal impairment will be enrolled. Two cohorts of 8 healthy participants will be enrolled. One cohort of healthy participants will be matched to the hepatic-impaired participants, whereas the other will be matched to the renal-impaired participants.

The study has 2 phases. The Pre-study Phase consists of a Screening Period and a Baseline Period. The Study Phase consists of a 2-day Study Period. No lenvatinib will be administered in this study.

The end of the study will be the date of the last study visit for the last participant in the study.

The following estimates are provided:

* From first participant in to last participant out, the study is expected to take approximately one year to complete.
* The maximum estimated duration of the study for each participant is anticipated to be approximately 5 weeks.

ELIGIBILITY:
Inclusion Criteria:

Key Inclusion Criteria:

* Male or Female
* Age, at the time of Informed Consent:

  i. Hepatic Impairment Participants (Including Matched Healthy Participants): 18 to 70 years old, inclusive ii. Renal Impairment Participants (Including Matched Healthy Participants): 18 to 79 years old, inclusive
* Non-smokers and smokers who smoke no more than 10 cigarettes per day
* Besides diabetes and, as appropriate, renal or hepatic impairment, participants must have no history of acute or chronic clinically relevant disease or condition, as determined by the investigator.
* For participants with hepatic impairment:

  * Liver cirrhosis that has been stable;
  * Platelet count >30,000 cells/millimeter cubed (mm^3);
  * Total score on the Child-Pugh classification system between 5 and 6 (Group 1, mild), 7 and 9 (Group 2, moderate), and 10 and 15 (Group 3, severe)
* For healthy participants:

  • Creatinine clearance ≥ 81 milliliter per minute (mL/min)
* For participants with renal impairment:

  * Must have a diagnosis of renal impairment that has been stable
  * Must have renal impairment in the following categories based on creatinine clearance values: mild (creatinine clearance, 50 to 80 mL/min), moderate (creatinine clearance, 30 to 49 mL/min), or severe (creatinine clearance, 15 to 29 mL/min) renal impairment

Exclusion Criteria:

Key Exclusion Criteria:

* Use of any new medication
* Human immunodeficiency virus (HIV) positive
* Presence of acute active liver disease or acute liver injury
* History of significant cardiovascular impairment
* Positive drug or alcohol test
* Weight loss or gain of >10% prior to Day 1
* Receipt of blood or blood products or donation of blood or blood products

For participants with hepatic impairment:

* History of hepatic transplant, systemic lupus erythematosus, or hepatic coma
* Received treatment with interferon or pegylated interferon
* Participants who have encephalopathy >Grade 2, sepsis, or gastrointestinal bleeding; esophageal varices >Grade 2, acute hepatic failure of any etiology, history of surgical portosystemic shunt, renal impairment (creatinine clearance <50 mL/min according to the Cockcroft-Gault formula), and rapidly deteriorating hepatic function
* Systolic blood pressure (SBP) ≥ 160 millimeters of mercury (mmHg) and/or diastolic blood pressure (DBP) ≥ 100 mmHg

For healthy participants:

• Hemoglobin level less than 12.0 grams per deciliter (g/dL)

For participants with renal impairment:

* A history of renal transplant
* SBP ≥ 160 mmHg and/or DBP ≥ 100 mmHg for participants with mild renal impairment; SBP ≥ 180 mmHg and/or DBP ≥ 110 mmHg for participants with moderate and severe renal impairment
* Significant bleeding diathesis

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2016-12-02 (Actual); Primary Completion 2017-07-08 (Actual); Study Completion 2017-07-08 (Actual)

PRIMARY OUTCOMES:
Number of participants with any serious adverse event and any non-serious adverse event | 1 week

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Orlando Clinical Research Center, Inc., Orlando, Florida
  - DaVita Clinical Research, Minneapolis, Minnesota
  - New Orleans Center for Clinical Research, Knoxville, Tennessee

IPD SHARING:
Plan to Share IPD: No